CLINICAL TRIAL: NCT04044781
Title: A Phase 1, Open-Label, Positron Emission Tomography Study in Healthy Subjects to Determine the Relationship Between Plasma Concentration and Brain Target Occupancy of BPN14770
Brief Title: A Phase 1, Open-Label, PET Study of T2310 & BPN14770
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Change in Research Direction
Sponsor: Tetra Discovery Partners (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: T2310-PET-102
Record Dates: First submitted 2019-08-02; First posted 2019-08-05 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: To Determine Brain Target Occupancy of BPN14770
MeSH Terms: interventions — BPN14770

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Test Group (Experimental): Stage 1 safety assessments will be performed before and after the administration of a single, 185 MBq (5mCi) dose of T2310 in up to three healthy volunteers. Stage 2 will evaluate the relationship between plasma concentration of BPN14770, an investigational PDE4D modulator, and brain target occupancy in up to six healthy volunteers.
  Interventions: Drug: BPN14770, T2310

INTERVENTIONS:
Drug: BPN14770, T2310 — Subjects will be administered radio ligand T2310 and BPN14770 to determine brain occupancy of BPN14770.

SUMMARY:
This is a sponsor initiated, single site, first-in-human study of an investigational imaging agent for quantifying the topographically specific concentrations of the phosphodiesterase enzyme Type 4D (PDE4D) with positron emission tomography (PET) using a selective radioligand, [11C]T2310. T2310 will be measured with imaging techniques to characterize plasma exposure levels versus regionally specific target engagement fractions for oral doses of BPN14770, an investigational new drug (IND) for modulating PDE4D. BPN14770 is under evaluation for the treatment of Fragile X syndrome and Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* 1. Willing and able to provide written informed consent.
* 2. Subjectively healthy
* 3. Between 18 and 75 years, inclusive, but preference will be given to subjects who are less than 55 years old.
* 4. The subject weighs at least 45 kg and has a body mass index between 18.0 and 32 kg/m2.
* 5. Subjects should be willing to observe the following contraception requirements from Screening until 90 days after the final follow-up visit: Male subjects must be willing to inform female partners of their participation in the study and must agree to use adequate contraceptive methods (vasectomy performed at least 6 months prior to dosing BPN14770 or use at least one barrier method of birth control). Female subjects: Female subjects must be surgically sterile (bilateral tubal ligation, hysterectomy, or bilateral oophorectomy at least 6 months prior to dosing of BPN14770), at least two years post-menopausal, or willing to use one barrier plus a hormonal contraceptive method of contraception from initial screening until one month after taking the last dose of study drug

Exclusion Criteria:

* 1. Known history or evidence of a clinically significant medical condition, disorder, or disease that, in the opinion of the investigator, would pose a risk to subject safety, proper completion of the procedures, or the integrity of the study.
* 2. Clinical laboratory studies suggestive of a medically meaningful disease or condition that, in the opinion of the investigator, could pose a risk to subject safety, proper completion of the procedures, or the integrity of the study.
* 3. Contraindication to MRI based on the standard MRI screening questionnaire at CBIC. Contraindications include ferromagnetic foreign bodies (e.g., shrapnel, ferromagnetic sheet metal fragments in the orbital area), certain implanted medical devices (e.g., older aneurysm clips, cardiac pacemakers), or claustrophobia.
* 4. Unexpected findings on screening MRI that are indicative of an occult brain disease, or will potentially compromise subject safety or the scientific integrity of the study data.
* 5. Previous exposure to ionizing radiation for research purposes, such that, in combination with the exposure from this study, their exposure to research associated radiation will be >50 mSv/year for the previous year.
* 6. Subjects who are atopic, or have a known hypersensitivity to any component of the formulation of BPN14770 or to [11C]T2310 PET scan.
* 7. History of substance dependence, or current use of drugs of abuse.
* 8. History of regular weekly alcohol consumption >21 units for male subjects or >14units for female subjects or unable to abstain from alcohol from 24 hours prior to Screening visits and 24 hours prior to Period 2 Day (-1) until discharge at the end of Period 2.

  9. Female subjects who are pregnant or lactating. 10. Use of any prescription drugs within 14 days or 5 half-lives (whichever is longer) before the first dose of an investigational product, unless in the opinion of the investigator (or delegate) and the Sponsor's Medical Monitor the medication will not interfere with the study procedures, the pharmacokinetics of either the radiopharmaceutical or the investigational drug product, or compromise subject safety. An example of potentially acceptable drug use might be beta blockers in eye drops for glaucoma.
* 11. Use of any non-prescription drugs, including vitamins, herbal and dietary supplements within 14 days or 5 half-lives (whichever is longer) before the first dose of the study agents, unless in the opinion of the Investigator (or delegate) and the Sponsor's Medical Monitor the medication will not interfere with the study procedures, the pharmacokinetics of either the radiopharmaceutical or the investigational drug product, or compromise subject safety.
* 12. Subjects who have received an investigational drug as part in another study within the last 30 days or 5 half-lives of the investigational drug for the previous study (whichever is longer).
* 13. History of acquired immunodeficiency syndrome (AIDS).
* 14. Poor peripheral venous access.
* 15. Donation of ≥450 mL blood or loss of blood during surgery within 30 days prior to Day 1.
* 16. Plasma donation >100 mL within 7 days prior to Day 1.
* 17. In the Investigator's judgement it is better for the subject not to be enrolled in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 1-8 Days
  To assess the safety and tolerability of [11C]T2310 when administered alone and when co-administered with BPN14770
Plasma Concentration | 24 Hours
  To determine relationships between plasma concentrations of BPN14770 and the total volume of distribution of T2310 as a proxy for brain PDE4D occupancy by BPN14770 following single oral dosing regimens of BPN14770 over a 24 hour time

CONTACTS AND LOCATIONS:
Overall Officials: Paul D Mozley, MD, Principal Investigator — Weill Cornell College of Medicine
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No